CLINICAL TRIAL: NCT02440893
Title: Understanding the Effect of Metformin on Corus CAD (MET Study)
Brief Title: Understanding the Effect of Metformin on Corus CAD (or ASGES)
Acronym: MET
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000018; MET Study (Other: CardioDx)
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CAD; CVD; CHD
Keywords: Corus CAD; ASGES; Age/Sex/Gene Expression Score; Gene Expression; GES; CAD; CVD; CHD; Precision Medicine; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; Metformin
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Corus CAD (ASGES) Post-metformin: Corus CAD (ASGES) second sample draw results to compare to Corus CAD (ASGES) first draw results (per patient).
  Interventions: Diagnostic Test: Corus CAD (ASGES)

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES)

SUMMARY:
The study goal was to understand the effect of Metformin on Age/Sex/Gene Expression Score (ASGES) or Corus CAD (henceforth "Corus") in pre-diabetic patients who are medication naive. This study provided data to determine if the Corus CAD (ASGES) signature was different in pre-diabetic patients when metformin was newly prescribed and taken.

DETAILED DESCRIPTION:
The study goal was to understand the effect of Metformin on Age/Sex/Gene Expression Score (ASGES) or Corus CAD in pre-diabetic patients who are medication naive. This study provided data to determine if the Corus CAD (ASGES) signature was different in pre-diabetic patients when metformin was newly prescribed and taken. The primary aim of this study was to evaluate whether metformin used in pre-diabetic patients to prevent progression to type II diabetes had a significant effect on the gene expression levels measured in Corus. This was a prospective study. Subjects were enrolled from participating sites as applicable inclusion/exclusion criteria were met. The study aimed to enroll approximately fifty (50) patients.

ELIGIBILITY:
Inclusion Criteria:

At least 21 years of age

Any of the following:

* Chest pain syndrome, stable angina, or anginal equivalent suggesting myocardial ischemia
* Low-risk unstable angina, or
* Asymptomatic individuals with a high probability of CAD

Clinician diagnosis of pre-diabetes, per ADA guidelines, such that metformin therapy is prescribed:

* HgA1C: >5.7% - <6.4%,
* BMI> 35 kg/m2
* Age< 60 yrs
* Prior Gestational Diabetes Mellitus
* FPG: >100mg/dl - <126mg/dl
* OGTT: >140mg/dl - <200mg/dl Willingness to comply with metformin therapy, for at least seven (7) days (P.O., per physician's dosage discretion) Willingness to maintain a drug diary for duration of study, for full follow-up period (7 + 7 days) Willingness and ability to provide two (2) samples for Corus (baseline, 7 (+ 7) days post- medication start) Provide written informed consent

Exclusion Criteria:

* History of or current level of HbA1C >6.5
* History of or current prescription of metformin or any other diabetic medication
* History of myocardial infarction (MI) or prior revascularization
* Current MI or acute coronary syndrome (ACS)
* Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms
* Current systemic infectious or systemic inflammatory conditions
* Subjects currently taking steroids, immunosuppressive agents or chemotherapeutic agents

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled from participating sites as applicable inclusion/exclusion criteria are met. The study aims to enroll approximately fifty (50) patients.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Metformin effect on Corus CAD | 7 days (+7days)
  Observe the effect of metformin use on Corus CAD (age, sex, gene expression score - ASGES) results

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mouton, MD, Principal Investigator — The Mouton Clinic